CLINICAL TRIAL: NCT00854204
Title: Phase I, Open-label, 3-way Crossover Trial in Healthy Male Volunteers to Evaluate the Pharmacokinetics of TMC114 and TMC41629 After a Single Oral Dose of 2 Controlled-release Coformulations as Compared to an Immediate-release Coformulation of TMC114/TMC41629
Brief Title: Innovation-TiFP4-C101: A Study to Evaluate the Pharmacokinetics of TMC114 and TMC41629 After a Single Oral Dose of 2 Controlled-release Coformulations as Compared to an Immediate-release Coformulation of TMC114/TMC41629
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015763
Record Dates: First submitted 2009-01-15; First posted 2009-03-03 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: HIV-I
Keywords: Innovation-TiFP4-C101; Innovation-C101; Innovation; TMC114/TMC41629; controlled-release coformulations; immediate-release coformulation; Pharmacokinetics
MeSH Terms: interventions — Darunavir

INTERVENTIONS:
Drug: TMC114; TMC41629

SUMMARY:
The purpose of this study is to compare the bioavailability (the degree to which a drug becomes available in the body after administration) of 3 different pharmaceutical preparations of a combination of two drugs, TMC114 and TMC41629. There will be 1 single oral intake (intake by mouth) of each of the 3 preparations. The study will also investigate the safety of use and the potential side effects of TMC114 and TMC41629, and determine the circulating levels of both compounds in your blood over time (pharmacokinetics), after a single intake.

DETAILED DESCRIPTION:
TMC41629 is a new investigational drug for the treatment of HIV. TMC114, is also known as Darunavir. In this randomized (study medication assigned by chance), open label trial (investigator and healthy volunteer know the name of the study medication), each healthy volunteer will receive a single dose of TMC114/TMC41629, in 3 subsequent sessions, Treatment A, Treatment B and Treatment C. Each capsule is equivalent to a dose of 200 mg of TMC114 and 23.67 mg of TMC41629. Treatment A (immediate-release formulation) will serve as reference formulation. All medication intakes will be orally and in fasted conditions.The study duration is at least 19 days, excluding screening and follow-up visits with three single intakes with 72 hours follow-up per intake. Each volunteer will receive a single dose of each formulation. TMC114/TMC41629 is formulated as an oral immediate-release hard-gelatin capsule, as an oral gastro-resistant hard-gelatin capsule, enteric-coated and as an oral gastro-resistant hard-gelatin capsule, colon-targeted. Each capsule is equivalent to a dose of 200 mg of TMC114 and 23.67 mg of TMC41629.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking for at least 3 months prior to selection
* Normal weight as defined by a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form (ICF) signed voluntarily before the first trial-related activity
* Able to comply with protocol requirements
* Healthy on the basis of a medical evaluation that confirms the absence of any clinically relevant abnormality and includes a physical examination, medical history, the results of blood biochemistry, coagulation, and hematology tests, a urinalysis, vital signs, and a 12-lead electrocardiogram (ECG) (in triplicate) with the following parameters carried out at screening: a. heart rate (HR) between 40 and 100 bpm
* b. QTc interval = 450 ms
* c. QRS interval lower than 120 ms
* d. PR interval = 220 ms.

Exclusion Criteria:

* Past history of heart arrhythmias
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the trial procedures
* Hepatitis A, B, or C infection or HIV-1 or HIV-2 infection at screening
* Currently active or underlying gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, endocrinologic, genitourinary, renal, hepatic, respiratory, inflammatory, or infectious disease
* Any history of significant skin disease and allergy to drugs

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Plasma levels of TMC114 and TMC41629 will be determined up to 72 hours after administration.

SECONDARY OUTCOMES:
To determine short-term safety and tolerability of TMC114/TMC41629 following administration of 3 single oral doses (formulated as different coformulations of TMC114/TMC41629).

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited